CLINICAL TRIAL: NCT06234488
Title: A Multi-Institutional Retrospect Cohort Study of Breast Cancer Diagnosis and Management in Transgender and Gender-Diverse Individuals
Brief Title: Multi-Institutional Transgender & Gender-Diverse Breast Cancer Study
Status: Active, not recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Chandler S Cortina, Assistant Professor of Surgery, Medical College of Wisconsin
Other Study IDs: PRO00043417
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Adenocarcinoma; Breast Cancer Stage; Breast Cancer Stage IV; Breast Cancer Invasive; Breast Cancer in Situ
Keywords: Transgender; Breast Cancer; Nonbinary; Gender Diverse; Gender-Affirming Hormone Therapy
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transgender and Gender-Diverse Persons with Breast Cancer: Patients who had a breast cancer diagnosis (including those with ductal carcinoma in situ (DCIS)), who were age ≥18 years at the time of diagnosis and identify as a gender and/or sex that is different from their sex assigned at birth (e.g., transgender, nonbinary, genderqueer, etc.) between 1/1/1990 - 7/1/2023.

SUMMARY:
There is no granular retrospective data on breast cancer in transgender and gender-diverse (TGD) persons from a contemporary and diverse American cohort. The purpose of this investigation is to aggregate data from multiple institutions to describe the risk, diagnosis, management, and outcomes of TGD persons with breast cancer in effort to identify opportunities for future intervention studies to eliminate breast cancer disparities for this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years of age or older
2. Breast cancer diagnosis (including DCIS)
3. Persons who identify as gender and/or sex that is different from the sex they were assigned at birth

Exclusion Criteria:

1. Age <18 at time of breast cancer diagnosis
2. Cis-gendered persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender and gender-diverse persons (TGD)
Study Population: Eligible patients are those who had a breast cancer diagnosis (including those with ductal carcinoma in situ (DCIS), who were age ≥18 years at the time of diagnosis and identify as a gender and/or sex that is different from the sex they were assigned at birth (e.g., transgender, nonbinary, genderqueer, etc.) between 1/1/1990 - 7/1/2023.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Breast Cancer Diagnosis Method | 33 years
  Describe the method of breast cancer diagnosis (self detected vs screen detected vs healthcare provider detected) and compare to the published data from cisgender women by determining means and standard deviation and comparing rates using the Wilcoxon signed-rank test.
Breast Cancer Risk Factors | 33 years
  Assess breast cancer risk factors (family history, genetics, etc.), including a prior use of gender-affirming hormone therapy and/or gender-affirming surgery on tumor receptor status and stage at diagnosis using t-test and chi-squared test.
Breast Cancer Management Strategies | 33 years
  Report breast cancer management strategies (type of breast surgery, receipt of radiation, etc.) through descriptive and comparative staststics with a focus on the use of adjuvant endocrine therapy and gender-affirming hormone therapy for patients with hormone-receptor positive disease using t-test and chi-squared test.
Outcomes Data | 33 years
  Breast cancer local and distant recurrence, overall survival, and disease-free survival using Kaplan-Meier analysis. Cox Proportional Hazards model will be used to estimate the effect of various factors on distant metastasis-free and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Chandler S Cortina, Principal Investigator — The Medical College of Wisconsin
Locations (22):
- United States (22):
  - University of Southern California/Los Angeles (USC/LA County), Los Angeles, California
  - University of California San Francisco (UCSF), San Francisco, California
  - University of Colorado Anschutz Medical Campus (CU Anschutz), Aurora, Colorado
  - MedStar Georgetown University Hospital (MGUH), Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center (MCC), Tampa, Florida
  - Northwestern Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Birgham and Women's Hospital, Boston, Massachusetts
  - Boston University (Boston U), Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - New York University (NYU), New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation (CCF), Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center (VUMC), Nashville, Tennessee
  - University of Washington (UW), Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin